CLINICAL TRIAL: NCT01768663
Title: A Phase 1, Open-Label Study to Examine the Effect of Ciprofloxacin, Itraconazole, and Rifampin on the Pharmacokinetics of Lumacaftor in Combination With Ivacaftor in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Examine the Drug-Drug Interaction of Ciprofloxacin, Itraconazole, and Rifampin on the Combination of Lumacaftor With Ivacaftor in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX12-809-009
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor; Ciprofloxacin; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Group (Cohort 1) (Experimental): Subjects will take lumacaftor in combination with ivacaftor for 14 days. Beginning on Day 15, subjects will take lumacaftor in combination with ivacaftor and ciprofloxacin through Day 21.
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor; Drug: Ciprofloxacin
- Treatment Group (Cohort 2) (Experimental): Subjects will take lumacaftor in combination with ivacaftor for 14 days. Beginning on Day 15, subjects will take lumacaftor in combination with ivacaftor and itraconazole through Day 21.
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor; Drug: Itraconazole
- Treatment Group (Cohort 3) (Experimental): Subjects will take lumacaftor in combination with ivacaftor for 14 days. Beginning on Day 15, subjects will take lumacaftor in combination with ivacaftor and rifampin through Day 24.
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor; Drug: Rifampin
- Treatment Group (Cohort 4) (Experimental): Subjects will take a single dose of lumacaftor in combination with ivacaftor on 3 occasions separated by 7 days.
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor

INTERVENTIONS:
Drug: Lumacaftor — tablet, 200mg taken every 12 hours
  Other Names: VX-809
Drug: Ivacaftor — tablet, 250mg taken every 12 hours
  Other Names: VX-770
Drug: Ciprofloxacin — 750 mg taken every 12 hours
  Arms: Treatment Group (Cohort 1)
Drug: Itraconazole — 200mg taken once daily
  Arms: Treatment Group (Cohort 2)
Drug: Rifampin — 600mg taken once daily
  Arms: Treatment Group (Cohort 3)

SUMMARY:
The purpose of this study is to examine the drug-drug interaction effects of ciprofloxacin, itraconazole, and rifampin on the pharmacokinetics of lumacaftor in combination with ivacaftor as well as to evaluate the potential effects of lumacaftor in combination with ivacaftor on lung function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects must be between the ages of 18 and 55 years, inclusive
* Body mass index (BMI) of 18 to 31 kg/m2, inclusive, and a total body weight >50 kg.

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject. This may include, but is not limited to, a history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; or history of mental disease.
* History of febrile illness within 5 days before the first dose.
* History of Gilbert's syndrome
* Abnormal renal function as defined at screening
* Blood donation of approximately 1 pint (500 mL) within 56 days before study drug administration
* Treatment with an investigational drug within 30 days or 5 half-lives (or as determined by the local requirements, whichever is longer) preceding the first dose of study drug
* Known hypersensitivity or prior adverse reaction to ciprofloxacin, or any member of the quinolone class of antimicrobial agents (Cohort 1 only); itraconazole, or to any of the other azoles (Cohort 2 only); rifampin, or to any of the rifamycins (Cohort 3 only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cohorts 1-3: PK parameters including Cmax, and AUC from time of dosing to time tau of lumacaftor and ivacaftor in the absence and presence of ciprofloxacin, itraconazole, and rifampin | up to 24 days
Cohort 4: Change in lung function from before treatment with lumacaftor/ivacaftor to after treatment with lumacaftor/ivacaftor. | up to 21 days

SECONDARY OUTCOMES:
Cohorts 1-4: Safety and tolerability as measured by adverse events (AEs) and changes in laboratory test values (serum chemistry, hematology, coagulation, and urinalysis), vital signs, standard 12 lead electrocardiograms (ECGs), and spirometry | up to 31 days
Cohort 4: PK parameters, including Cmax of lumacaftor/ivacaftor, and lung function | 16 days

CONTACTS AND LOCATIONS:
Locations (1):
- Evansville, Indiana, United States